CLINICAL TRIAL: NCT03453814
Title: Music Intervention for Agitation Reduction in the Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, David Rothstein, Associate Professor of Surgery, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001771
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Critical Illness
Keywords: PICU; critical care; music; music therapy; agitation
MeSH Terms: conditions — Critical Illness; Psychomotor Agitation | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Music therapy.
  Interventions: Other: Music Therapy
- Comparison (No Intervention): No music therapy.

INTERVENTIONS:
Other: Music Therapy — Subjects will receive one hour of music twice a day for three days.
  Arms: Interventional

SUMMARY:
The objective of this study is to administer music therapy to patients in the pediatric intensive care unit (PICU) in order to observe how music affects patient agitation, vital signs, and overall recovery in the unit.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled study to observe patients who have been admitted to the PICU with an altered state of agitation according to the Richmond Agitation Sedation Scale (RASS). These patients will be administered music therapy during a controlled setting in the day to observe whether the introduction of music therapy helps reduce the patient's level of agitation, improving their vital signs and overall recovery in the unit. Once patients are enrolled and have signed consents, patients will receive a headset with music or dead air. Therapy times will be selected so that there are minimal disruptions. Total time will be 2 hours daily, once in the morning and once in the evening. The treatments for session 1 and session 2 of the day will be the same (i.e. Music/ Music, No music/No Music).

The investigators hypothesize that applying music therapy in the PICU will decrease agitation, length of stay, and narcotic administration, and normalize heart rate, respiratory rate, and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* PICU patient at Oishei Children's Hospital of Buffalo
* >4 years of age, <18 years of age
* Patients with RASS of +1

Exclusion Criteria:

* Documented underlying psychological disorders
* Diagnosed with sever developmental delay
* Prior narcotic dependence
* Underlying medical conditions affecting heart rate, blood pressure, or neuromuscular system
* Chemically paralyzed patients
* Anyone with an aneurysm
* Patients who are deaf in both ears
* Ear bone fractures or other middle/inner ear trauma or major ear avulsion as determined by physician
* Hemodynamically unstable patients
* Patients facing imminent death

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Richmond Agitation-Sedation Scale (RASS) | 3 days
  The Richmond Agitation-Sedation Scale (RASS) is a medical scale used to measure the agitation or sedation level of a patient. The scale measures patient agitation and sedation +4 to -5, with a score of 0 equal to an alert and calm patient, a positive score equal to various levels of aggression, and a negative score equal to various levels of sedation. Patients receive one score for one observed time point. Therefore, a patient will have one score from +4 to -5. For the purpose of this study, a better outcome will be a score that is around 0 or that decreases from a higher positive score to a lower positive score. The investigators hypothesize that music therapy will decrease agitation in patients and decrease their positive RASS score.

SECONDARY OUTCOMES:
Bispectral Index (BIS) | 3 days
  The Bispectral Index provides a direct measure of the effects of sedatives on the brain. It is an algorithm developed by Aspect Medical Systems that measures EEG after the administration of anesthetic agents and is measure on a BIS monitor. The BIS monitor reports a single number from 0 to 100 that represents an integrated measure of cerebral electrical activity. This is interpreted into a patient's level of alertness. A score of 100 indicates that the patient is fully awake, while a number less than 40 is suggestive of a deep hypnotic effect. For the purpose of this study, the investigators are using the BIS to measure the level of alertness in a patient. The investigators hypothesize that the administration of music therapy with have a sedative effect on patients, thereby decreasing their BIS number.

CONTACTS AND LOCATIONS:
Overall Officials: David Rothstein, MD, Principal Investigator — SUNY Buffalo
Locations (1):
- Oishei Children's Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kudchadkar SR, Berger J, Patel R, Barnes S, Twose C, Walker T, Mitchell R, Song J, Anton B, Punjabi NM. Non-pharmacological interventions for sleep promotion in hospitalized children. Cochrane Database Syst Rev. 2022 Jun 15;6(6):CD012908. doi: 10.1002/14651858.CD012908.pub2. PMID 35703367